CLINICAL TRIAL: NCT00076349
Title: A Multi-Center Phase II Study to Investigate the Safety and Activity of SDX-105 (Bendamustine) in Combination With Rituximab in Patients With Relapsed Indolent or Mantle Cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: SDX-105 in Combination With Rituxan for Patients With Relapsed Indolent or Mantle Cell Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDX-105-02
Record Dates: First submitted 2004-01-20; First posted 2004-01-22 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; NHL; Rituxan; Mantle Cell; mabs
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride; Rituximab

ARMS (1):
- 1 (Experimental): open-label, single arm, clinical trial of bendamustine (SDX-105) plus rituximab
  Interventions: Drug: bendamustine and rituximab

INTERVENTIONS:
Drug: bendamustine and rituximab — Patients will receive rituximab on the first day of a cycle at a dose of 375 mg/m2, followed on the second and third day of a cycle by SDX-105 (bendamustine) at a dose of 90 mg/m2/day of treatment. Four cycles are planned. Patients will receive a dose of rituximab alone 7 days prior to the first cycle of the combination and a dose of rituximab 28 days after the last cycle of the combination. If there is documented disease regression, a fifth and sixth cycle of SDX-105 plus rituximab may be administered.

SUMMARY:
SUMMARY:

This is an open label study combining Rituxan and SDX-105. Rituxan will be given on day 1 followed by a 30-60 minute intravenous infusion of SDX-105 on day 2 and day 3. Treatment will repeat every 21 days (a cycle). Treatment can continue for up to 6 cycles (about 4 months) if tumor status improves and there are no unacceptable side effects. Patients will be followed for up to 2 years or until disease progression.

RATIONALE:

Rituxan has been shown to increase the sensitivity of cells to chemotherapy. The combination of SDX-105 and Rituxan has been effective in both the laboratory and in a recent clinical study with Non-Hodgkin's lymphoma patients.

PURPOSE:

This study will evaluate the safety and effectiveness of SDX-105 plus Rituxan in patients with Non-Hodgkin's lymphoma who have relapsed after taking Rituxan.

ELIGIBILITY:
INCLUSION CRITERIA:

Documented B-Cell NHL or mantle cell lymphoma

* CD-20+ tumor
* Indolent NHL: follicular B-cell lymphoma, diffuse small lymphoma, marginal zone lymphoma
* Maximum of three prior chemotherapy regimens
* Age of at least 18 years at Screening Visit (Site specific requirement may differ)

EXCLUSION CRITERIA:

* Refractory to rituximab, defined as progression of disease while being treated with rituximab or progression within 6 months of the last dose of rituximab (when given either as a single agent or in combination)
* Previous chemotherapy or immunotherapy within 3 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin) or failure to recover from adverse events due to any agents administered previously
* Use of investigational agents within 28 days of study
* History of prior high dose chemotherapy with allogeneic stem cell support
* History of prior radioimmunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2004-04; Primary Completion 2005-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Determine the objective response rate (ORR = CR + PR) to a regimen of SDX-105 plus rituximab in patients with relapsed indolent or mantle cell non-Hodgkin's lymphoma | 4-6 months

SECONDARY OUTCOMES:
• To characterize the safety profile of SDX-105 plus rituximab in this patient population • To determine the one-year and Kaplan-Meier estimates of progression-free survival (PFS) rates • To determine the median duration of response (DR) | 4-6 months

CONTACTS AND LOCATIONS:
Locations (34):
- United States (25):
  - Alaska Cancer Research and Education Center, Anchorage, Alaska
  - Bay Area Cancer Research Group, Concord, California
  - Wilshire Oncology Medical Group, La Verne, California
  - USC/Kenneth Norris Jr. Cancer Hospital and Research Institute, Los Angeles, California
  - San Diego Cancer Center, Vista, California
  - Hematology Oncology, P.C. Carl and Dorothy Bennett Cancer Center, Stamford, Connecticut
  - Georgetown University Medical Center - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Pasco Hernando Oncology, New Port Richey, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Suburban Hematology & Oncology Associates, Lawrenceville, Georgia
  - Georgia Oncology Partners Research and Education Foundation, Macon, Georgia
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Oncology and Hematology, Metairie, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Beth Israel/Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Arena Oncology Associates, Great Neck, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Upstate NY Cancer Research & Education Foundation, Inc. - Interlakes Oncology/Hematology, Rochester, New York
  - ACORN - West Cancer Center, Memphis, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Univ. of Virginia Health System-Cancer Center Clinical Trials Office, Charlottesville, Virginia
- Australia (4):
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - St. Vincent's Hospital, Darlinghurst
  - Westmead Hospital, Westmead
- Canada (5):
  - Queen Elizabeth II Health Sciences Centre-Victoria General Site, Halifax, Nova Scotia
  - The Royal Victoria Hospital Cancer Care Program Clinical Trials, Barrie, Ontario
  - North Eastern Ontario Regional Cancer Center, Greater Sudbury, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Hopital Notre-Dame Du Chum, Montreal, Quebec